CLINICAL TRIAL: NCT06471634
Title: An Efficacy Study Exploring the Optimisation of Sleep and the Reduction of Sedentary Behaviour in Those Living With Type 2 Diabetes Mellitus
Brief Title: A Study Looking to Improve Sleep and Reduce Sedentary Behaviour in Those Living With Type 2 Diabetes Mellitus
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leicester (Other)
Collaborators: University Hospitals, Leicester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0955; 334347 (Other: IRAS)
Record Dates: First submitted 2024-06-10; First posted 2024-06-24 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Diabetes Mellitus, Type 2; Insomnia; Sedentary Behavior
Keywords: Sleep; Insomnia; Sedentary behaviour; Diabetes Mellitus, Type 2; Cognitive Behaviour Therapy insomnia (CBTi); Behaviour change
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Sleep Initiation and Maintenance Disorders; Sedentary Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The technicians analysing the accelerometer data and blood analysis will be blinded as to which arm the participant is from, no other masking is possible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBTi and Sedentary Behaviour support (Experimental): Participants will be counselled in how to improve their sleep and decrease sedentary behaviour using CBTi and behaviour change techniques.
  Interventions: Behavioral: CBTi; Behavioral: Sedentary behaviour reduction
- Control - usual care (Active Comparator): Participants will be given a leaflet containing brief information on good sleep hygiene practice and the benefits of decreasing sedentary behaviour.
  Interventions: Other: Control - usual care

INTERVENTIONS:
Behavioral: CBTi — A 12 week intervention using CBTi to improve sleep measured using objective and subjective measures. Participants will complete a number of questionnaires and tests at baseline and at completion to allow comparisons to be made.
  Arms: CBTi and Sedentary Behaviour support
Other: Control - usual care — Participants will be given a leaflet summarising good sleep practice and the advantages of reducing sedentary behaviour. Participants will complete a number of questionnaires and tests at baseline and at completion to allow comparisons to be made.
  Arms: Control - usual care
Behavioral: Sedentary behaviour reduction — Participants will be encouraged to increase activity and thus reduce sedentary time. Investigators will use behaviour change techniques to aid in this goal. Participants will complete a number of questionnaires and tests at baseline and at completion to allow comparisons to be made.
  Arms: CBTi and Sedentary Behaviour support

SUMMARY:
The goal of this clinical feasibility trial is to learn whether the investigators can improve sleep and reduce sedentary behaviour in people living with Type 2 diabetes mellitus with sleep problems. The main questions it aims to answer are: • question 1, can objectively measured sleep and sedentary behaviour be improved in the participants and • question 2, what effect will this have on a number of physical and physiological markers. Participants in the intervention group will be asked to keep sleep diaries and attend regular meetings with a qualified coach who will use a specific talking therapy to try to improve sleep and with use behaviour change techniques to help them be less sedentary. Researchers will compare the control group to the intervention group to see if effects differ between groups.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Diabetes Mellitus type 2 for longer than 3 months
* Participant is willing and able to give informed consent to take part in the study.
* Sleep disorder symptom checklist 25 (SDS-CL-25) of ≥5 on insomnia criteria.
* Not at high risk of undiagnosed Obstructive Sleep Apnoea (OSA), scoring ≥5 on STOP BANG scale (snoring, tired, observed, pressure, body mass index, age, neck size, gender) diagnosed treated OSA is acceptable.
* Glycated haemoglobin (HbA1c) of 10% or less (86 mmol/mol) or less
* Male or Females.
* ≥ 18 ≤ 75 years of age.
* Able to walk without the use of an assistive device or requiring assistance from another person.
* Not undertaking more than 75 minutes a week of strenuous exercise or sport.
* Not taking opioids
* Be treatment stable for at least 3 months
* Accelerometer measurement of SE ≤ 85%
* An understanding that CBTi may exacerbate sleep deprivation in the short term which may impact on certain aspects of daily life.

Exclusion Criteria:

* Individuals living with narcolepsy or diagnosed parasomnia
* Individuals with type 1 diabetes or gestational diabetes
* Recent cardiovascular event (within the last 6 months).
* Currently on opioids
* Diagnosed with borderline personality disorder, psychosis, adult attention deficit hyperactivity disorder (ADHD) or schizophrenia (self-reported).
* Individuals living with epilepsy or seizures.
* Shift workers
* Female participant planning to become pregnant with the timeframe of the study or is currently pregnant.
* Terminal illness.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-09-02 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Sleep Efficiency (SE) measured using accelerometer data. | Before and after the 12 week intervention/intervention period
  The primary outcome measure is change in objectively measured SE in the intervention arm compared to the control group.

SECONDARY OUTCOMES:
Objectively measured sleep - sleep onset latency | Before and after the 12 week intervention/intervention period
  Accelerometer data will be used to measure sleep onset latency in minutes.
Objectively measured sleep - wake after sleep onset | Before and after the 12 week intervention/intervention period
  Accelerometer data will be used to measure wake after sleep onset in minutes.
Objectively measured sleep - total sleep time | Before and after the 12 week intervention/intervention period
  Accelerometer data will be used to measure total sleep time in minutes.
Objectively measured sleep - sleep duration variability | Before and after the 12 week intervention/intervention period
  Accelerometer data will be used to measure sleep duration variability in minutes.
Objectively measured sleep - sleep midpoint variability | Before and after the 12 week intervention/intervention period
  Accelerometer data will be used to measure sleep midpoint variability in minutes.
Objectively measured sedentary behaviour | Before and after the 12 week intervention/intervention period
  Accelerometer data will be used to measure total time spent in sedentary time in minutes.
Objectively measured physical activity | Before and after the 12 week intervention/intervention period
  Accelerometer data will be used to measure total time spent in physical activity in minutes.
Subjectively measured sleep - insomnia | Before and after the 12 week intervention/intervention period
  The Insomnia Severity index, will be used to measure the level of insomnia - it is a questionnaire and has a range of 0-28 with higher scores indicating more insomnia.
Subjectively measured sleep quality - | Before and after the 12 week intervention/intervention period
  The Pittsburgh Sleep Quality Index will be used to measure subjective sleep quality, this is a questionnaire and has a range of 0-21 with higher scores indicating worse sleep quality.
Subjectively measured sleepiness | Before and after the 12 week intervention/intervention period
  Epworth Sleepiness Scale is a questionnaire and has a range of 0-24 with higher scores indicating more sleepiness.
Measurement of fatigue | Before and after the 12 week intervention/intervention period
  The Functional assessment of chronic illness therapy (FACIT) scale will be used to subjectively measure fatigue, the range is 0-52 with higher scores indicating less fatigue.
Blood pressure | Before and after the 12 week intervention/intervention period
  Blood pressure (both diastolic and systolic) will be measured using an automatic electronic device and the units used will be millimetres of mercury.
Fasting blood glucose | Before and after the 12 week intervention/intervention period
  Fasting measured via a venous sample and in millimoles per litre (Mmol/L)
Continuous blood glucose | Before and after the 12 week intervention/intervention period
  Continuous blood glucose measured via a continuous glucose monitor and in Mmol/L (Mmol/L)
Insulin | Before and after the 12 week intervention/intervention period
  Insulin will be measured via a venous sample and in micro units per millilitre.
Triglycerides | Before and after the 12 week intervention/intervention period
  Triglycerides will be measured via a venous sample and in Mmol/L.
Cholesterol | Before and after the 12 week intervention/intervention period
  Cholesterol, including Low density lipoprotein and high density lipoprotein and total cholesterol, will be measured via a venous sample and in Mmol/L
Physical function - the short physical performance battery | Before and after the 12 week intervention/intervention period
  The short physical performance battery consists of 3 physical tests, with a total score range of 0-12 with higher scores indicating better physical function.
Physical function - the sit to stand-60 | Before and after the 12 week intervention/intervention period
  The sit to stand-60 is the number of times the participant can rise from sit to stand in one minute using a designated chair with no arms and without the use of the participants arms, and is reported as a number.
Physical and Cognitive function - The World Health Organisation Disability Assessment schedule (WHODAS) | Before and after the 12 week intervention/intervention period
  WHODAS is a questionnaire used to assess both physical and cognitive function. Each question is scored 0-4, scores are then averaged for all the questions so the range is 0-4 and the higher the score the more difficulty the participant is experiencing in functioning.
Cognitive function - verbal fluency test | Before and after the 12 week intervention/intervention period
  Cognitive function will be measured using the verbal fluency test, which is conducted over two 60s periods and is scored by the number of correct answers.
Quality of life- European Quality of Life 5 dimension (EQ-5D-5L) | Before and after the 12 week intervention/intervention period
  EQ-5D-5L, the five questions are scored 1-5 and each represents a different aspect, it is presented as a five digit number representing each domain. The higher the numbers, the worse quality of life.
Weight | Before and after the 12 week intervention/intervention period
  Weight in kilograms will be measured.
Height | Before and after the 12 week intervention/intervention period
  Height in metres will be measured.
Body mass index (BMI) | Before and after the 12 week intervention/intervention period
  BMI will be calculated using weight and height to produce BMI in kg/m^2
Body composition - via bioimpedance | Before and after the 12 week intervention/intervention period
  Bioimpedance scales will be used to measure body composition including percentage fat, muscle mass and water
Depression - The Patient Health Questionnaire-9 (PHQ9) | Before and after the 12 week intervention/intervention period
  PHQ9 will be used to measure depressive symptoms. The PHQ9 has a range of 0-27 with higher scores indicating more depressive symptoms/depression.
Anxiety - The General Anxiety Disorder Assessment-7 (GAD7) | Before and after the 12 week intervention/intervention period
  GAD7 will be used to measure anxiety symptoms. It has a range of 0-21, with higher scores indicating more anxiety.
Food intake - food diaries | Before and after the 12 week intervention/intervention period
  3 Day food diaries will be used to measure food intake.

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Davies, PhD, Principal Investigator — Leicester Diabetes Centre
Locations (1):
- Diabetes Research Centre University Hospitals Leicester, Leicester, Leicestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Data in anonymised form may be suitable for sharing at the end of the trial. Should there be concerns about protecting the identity of participants/commercialisation of outputs, access restrictions will need to be considered. If suitable, anonymised data may be added to UoL's Research Archive (https://figshare.le.ac.uk/) within 6 months of the trial end date. The repository is registered in OpenDOAR and preserves research outputs (minimum of 10 years).